CLINICAL TRIAL: NCT05189197
Title: Efficacy and Safety of Zanubrutinib in Combination With R-CHOP in Newly Diagnosed Non-GCB DLBCL Patients With Double Expression: A Single-arm, Open-label, Phase II Study
Brief Title: A Study to Evaluate Efficacy and Safety of Zanubrutinib With R-CHOP in Newly Diagnosed Non-GCB DLBCL Patients With Double Expression
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Baotou Cancer Hospital (Other); Xiangya Hospital of Central South University (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Junning Cao, MD, Chief of department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRCHOP-BGB-3111-2004-IIT
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B-cell Lymphoma(DLBCL)
Keywords: Diffuse large B-cell lymphoma; Zanubrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Zanubrutinib + R-CHOP (Experimental): Zanubrutinib 160 mg bis in die（BID） administered by oral every day of each 21-day cycle. Rituximab 375 mg/m2, Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 (maximum total 2 mg) administered by IV infusion on Day 1 of each 21-day cycle.
  Prednisone 100 mg administered by oral on Day 1-5 of each 21-day cycle. After 6 cycles of zanubrutinib and R-CHOP combination therapy, patients achieved complete response （CR）will continue to receive zanubrutinib 160mg BID for 1 year.
  Interventions: Drug: Zanubrutinib + R-CHOP

INTERVENTIONS:
Drug: Zanubrutinib + R-CHOP — Zanubrutinib 160 mg BID administered by oral every day of each 21-day cycle. Rituximab 375 mg/m2, Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 (maximum total 2 mg) administered by IV infusion on Day 1 of each 21-day cycle.
  Prednisone 100 mg administered by oral on Day 1-5 of each 21-day cycle. After 6 cycles of zanubrutinib and R-CHOP combination therapy, patients achieved CR will continue to receive zanubrutinib 160mg BID for 1 year.
  Other Names: Brukinsa+Mabthera +CHOP

SUMMARY:
Zanubrutinib is a highly specific, potent new Bruton's tyrosine kinase （BTK） inhibitor, with minimal off-target inhibition of other kinases. This is a single-arm, open-label Phase II study to evaluate the efficacy and safety of zanubrutinib in combination with Rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in newly diagnosed non-GCB Diffuse large B-cell lymphoma (DLBCL) patients with co-expression of B-cell lymphoma 2 （BCL2）and myelocytomatosis oncogene（MYC）.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma as the most common lymphoma, is heterogeneous. R-CHOP is the standard care in front-line DLBCL treatment. However, there are still about 40% of the DLBCL patients treated with R-CHOP relapse or respond poorly.

There are 20%-30% DLBCL patients having BCL2 and MYC co-expression, which are more common in activated B -cell-like（ABC）-DLBCL. Previous study showed that patients with co-expression of BCL2 and MYC by immunohistochemistry (IHC) have a worse outcome with R-CHOP.

Efficacy results from Studies PCYC-04753 and PCYC-1106-CA demonstrate that BTK inhibitor ibrutinib has some activity as a single agent in subjects with relapsed or refractory DLBCL, with possible lower response rates in subjects with the germinal center B-cell-like （GCB）subtype.

In post hoc of PHEONIX study, non-GCB subgroup pts with MYC-high + BCL2-high had better event free survival （EFS ）(HR 0.648; 95% confidence interval （CI), 0.423-0.993; p = 0.045) with ibrutinib + R-CHOP versus placebo + R-CHOP.

Zanubrutinib is a highly specific, potent new BTK inhibitor, with minimal off-target inhibition of other kinases, and is associated with better tolerability, compared with ibrutinib. A post hoc analysis on 4 studies found that Patients with MYC and BCL2 double-expressor DLBCL resulted in objective response rate（ORR）of 61% and progression free survival (PFS) of 5.4m when treated with zanubrutinib. However, it is still unknown the benefit of zanubrutinib and RCHOP combination therapy followed by zanubrutinib maintenance in non-GCB DLBCL patients with co-expression of BCL2 and MYC.

This is a single-arm, phase II study, to evaluate the efficacy and safety of zanubrutinib in combination with R-CHOP followed by zanubrutinib maintenance in newly diagnosed non-GCB subtype of DLBCL patients with MYC-high + BCL2-high selected by IHC.

The study will include a Screening Phase, Combination Treatment Phase, Maintenance phase and a Post Treatment Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* No prior treatment for DLBCL.
* Histologically - confirmed non-GCB subtype.
* MYC+≥40% and BCL2+≥50% by IHC
* Lesions must be measurable. A measurable node lesion must have a longest diameter greater than 1.5 cm. A measurable extra-nodal lesion should have a longest diameter greater than 1.0 cm.
* Eastern Cooperative Oncology Group performance status grade of 0, 1, or 2
* Stage II (not candidates for local X-ray therapy), III, or IV disease by the Ann Arbor Classification
* Hematology values must be within the following limits at baseline:

  * Neutrophils ≥ 1 x 109/L, independent of growth factor support within 7 days of initiation of the combination therapy.
  * Platelets ≥ 75x 109/L, independent of growth factor support or transfusion within 7 days of initiation of the combination therapy. (platelets≥ 50 x 109/L, if there is bone marrow involvement.)
* Biochemical values must be within the following limits at baseline:

  * Alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN). Aspartate aminotransferase (AST) ≤3 x ULN.
  * Total bilirubin ≤1.5 x ULN, unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
  * Serum creatinine ≤2 x ULN or estimated Glomerular Filtration Rate≥40 mL/min/1.73m2
* International normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5 x ULN.

Able to provide written informed consent, can understand and comply breastfeeding are ineligible for this study.

Exclusion Criteria:

* Primary mediastinal lymphoma.
* Central nervous system involvement lymphoma.
* Histologically transformed lymphoma.
* Diagnosed or treated for malignancies other than DLBCL.
* History of stroke or intracranial hemorrhage within 6 months.
* Major surgery within 4 weeks.
* Required ongoing treatment with medication that are strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or strong/median effect CYP3A inducers.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification, or Echocardiography: Left ventricular ejection fraction (LVEF) < 50%
* Active, clinically significant Electrocardiogram (ECG) abnormalities including second degree atrioventricular (AV) block Type II, or third-degree AV block or QT interval corrected for heart rate (QTcF) prolongation, defined as a QTcF > 450 msec.
* Any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Known human immunodeficiency virus (HIV) infection, or active hepatitis B or hepatitis C infection.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of zanubrutinib capsules, or put the study outcomes at undue risk.

Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
3-year event-free survival (EFS) rate | up to 3 years
  3-year EFS rate is defined as the proportion of patients free from EFS events at 3 years after the initiation of zanubrutinib and RCHOP combination therapy estimated using the Kaplan-Meier method. EFS is defined as the duration from the initiation of zanubrutinib and RCHOP combination therapy to the date of documented disease progression, relapse from CR, initiation of subsequent systemic anti-lymphoma therapy for either positron emission computed tomography (PET)-positive or biopsy-proven residual disease after six cycles of Zanubrutinib and R-CHOP combination therapy, or any-cause death whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 18 weeks
  ORR is defined as the proportion of patients achieving complete response (CR) and partial response (PR), as per Lugano Classification.
Complete response rate (CRR) | up to 18 weeks
  CRR is defined as proportion of patients achieving CR, as determined per Lugano Classification.
3-year progression-free survival rate （PFS) | up to 3 years
  3-year PFS rate is defined as the proportion of patients free from PFS events at 3 years after the initiation of zanubrutinib and RCHOP combination therapy estimated using the Kaplan-Meier method. PFS is defined as the duration from the initiation of zanubrutinib and RCHOP combination therapy to the date of disease progression, relapse from CR, or death, whichever occurs first.
3-year overall survival (OS) rate | up to 3 years
  3-year OS rate is defined as the proportion of patients alive at 3 years after the initiation of zanubrutinib and RCHOP combination therapy estimated using the Kaplan-Meier method. OS is defined as the duration from the date of initiation of zanubrutinib and RCHOP combination therapy to the date of death.
adverse event（AE） | up to 2 years
  The incidence and severity of treatment-emergent adverse events (TEAEs), serious adverse event（SAEs）and reatment-related AEs according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No